CLINICAL TRIAL: NCT03539003
Title: The Comparison of Changes of QTc, Tp-e Interval, and Tp-e/QT Ratio, Tp-e/QTc Ratio on the ECG During Robotic-assisted Laparoscopic Radical Prostatectomy Under Sevoflurane, Desflurane and Total Intravenous Anesthesia -Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2018-0296
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Robotic-assisted Laparoscopic Radical Prostatectomy
MeSH Terms: interventions — Sevoflurane; Desflurane; Propofol; Remifentanil; Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: 1. sevoflurane group
  2. desflurane group
  3. total intravenous anesthesia group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sevoflurane (Group S) (Experimental): general anesthesia with sevoflurane
  Interventions: Drug: sevoflurane
- desflurane (Group D) (Active Comparator): general anesthesia with desflurane
  Interventions: Drug: desflurane
- total intravenous anesthesia (Group T) (Active Comparator): general anesthesia with total intravenous anesthesia
  Interventions: Drug: propofol and remifentanil

INTERVENTIONS:
Drug: sevoflurane — anesthesia was induced with propofol (1.5 mg/kg) and target controlled infusion (TCI) of remifentanil (2-3 ng/mL of targeted effect site concentration (Ce). After intubation, inspired concentration of sevoflurane (0.8-1 MAC) and the Ce of remifentanil TCI (1.0-2.0 ng/ml) were adjusted to a BIS target level for hypnosis of 40-60 during surgery.
  Other Names: Group S
  Arms: sevoflurane (Group S)
Drug: desflurane — anesthesia was induced with propofol (1.5 mg/kg) and target controlled infusion (TCI) of remifentanil (2-3 ng/mL of targeted effect site concentration (Ce). After intubation, inspired concentration of desflurane (0.8-1 MAC) and the Ce of remifentanil TCI (1.0-2.0 ng/ml) were adjusted to a BIS target level for hypnosis of 40-60 during surgery.
  Other Names: Group D
  Arms: desflurane (Group D)
Drug: propofol and remifentanil — anesthesia was induced with an effect-site concentration of 3-4 μg/ml propofol and 2-3 ng/ml remifentanil using target-controlled infusion (TCI). After intubation, The effect site TCI of propofol (2-3 μg/ml) and remifentanil (1.0-2.0 ng/ml) was adjusted to maintain the desired hypnosis (40-60 of the BIS value) during surgery.
  Other Names: Group T
  Arms: total intravenous anesthesia (Group T)

SUMMARY:
The purpose of this study is to compare the changes of QTc, Tp-e interval, and Tp-e/QT ratio, Tp-e/QTc ratio on the ECG during robotic-assisted laparoscopic radical prostatectomy under sevoflurane, desflurane and total intravenous anesthesia

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I-III
2. patients undergoing elective robot-assisted laparoscopic radical prostatectomy
3. adult (≥19 years old)

Exclusion Criteria:

1. emergency surgery
2. preoperative QTc prolongation
3. Cardiac disease (unstable angina, congestive heart failure, valvular heart disease)
4. uncontrolled hypertension (DBP >110 mmHg)
5. Patients who take beta blocker
6. Ventricular conduction abnormality
7. Hepatic or renal failure
8. Drug hyperactivity
9. patients unable to understand informed consent (foreigner, illiteracy..)

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients undergoing robotic-assisted laparoscopic radical prostatectomy
Enrollment: 69 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
heart-rate corrected QT(QTc) interval | participants will be followed for the duration of surgery, an expected average of 4 hours.
  QTc intervals (msec) are recorded from ECG

SECONDARY OUTCOMES:
Tp-e interval | Baseline (T0), 10 min after induction (T1), 5, 15, 30, 45, 60 min after Trendelenburg position (T2-6), 5 min after desufflation and resuming the supine position (T7), end of surgery (T8)
Tp-e/QT ratio | Baseline (T0), 10 min after induction (T1), 5, 15, 30, 45, 60 min after Trendelenburg position (T2-6), 5 min after desufflation and resuming the supine position (T7), end of surgery (T8)
Tp-e/QTc ratio | Baseline (T0), 10 min after induction (T1), 5, 15, 30, 45, 60 min after Trendelenburg position (T2-6), 5 min after desufflation and resuming the supine position (T7), end of surgery (T8)
Heart rate | Baseline (T0), 10 min after induction (T1), 5, 15, 30, 45, 60 min after Trendelenburg position (T2-6), 5 min after desufflation and resuming the supine position (T7), end of surgery (T8)
blood pressure | Baseline (T0), 10 min after induction (T1), 5, 15, 30, 45, 60 min after Trendelenburg position (T2-6), 5 min after desufflation and resuming the supine position (T7), end of surgery (T8)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No